CLINICAL TRIAL: NCT03781024
Title: The Purpose of This Study is to Evaluate the Level of Relief Perceived by Patients Using Medicated Footbath/Footwash With or Without an Oral Medication for the Treatment of: Toenail Fungus Ingrown Toenails Cellulitis Athletes' Foot Pitted Keratolysis Diabetic Ulcers Open Infected Sores Abscesses Joint Infections Wound Care
Brief Title: A Subjective Observational Study of Patients Using Medicated Footbath/Footwash Treatment in Podiatry Care
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Data Collection Analysis Business Management (Other)
Responsible Party: Sponsor
Other Study IDs: PAS1467
Record Dates: First submitted 2018-12-18; First posted 2018-12-19 (Actual); Last update posted 2018-12-19 (Actual); Status verified 2018-12

CONDITIONS: Toenail Fungal Infection; Cellulitis; Pitted Keratolysis; Diabetic Foot Ulcer; Abscess
MeSH Terms: conditions — Cellulitis; Diabetic Foot; Abscess

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Combination Product: Footwash — footbath/footwash can help cleanse the wound, remove dead tissue, increase circulation and puts the wound in direct contact with medication to promote faster healing.
  Other Names: Footbath

SUMMARY:
The purpose of this study is to evaluate the level of relief perceived by patients using medicated footbath/footwash with or without an oral medication for the treatment of podiatry issues.

DETAILED DESCRIPTION:
Footwash/Footbath for treatment of; Toenail fungus Ingrown toenails Cellulitis Athletes' foot Pitted Keratolysis Diabetic ulcers Open infected sores Abscesses Joint infections Wound care

ELIGIBILITY:
Inclusion Criteria:

Participants must be diagnosed with an ICD10 code indicative of Toenail Fungus, Ingrown Toenail, Cellulitis, Athletes Foot, Pitted Keratolysis, Diabetic Ulcers, Open infected sores, Abscesses, and Joint infections

* Participants must be starting a new regimen of a medicated footwash/foothbath
* Participants must be expecting to receive therapy for at least 12 weeks
* Participants must be between 18 and 64 years of age
* Participants must be able to provide sound verbal informed consent

Exclusion Criteria:

-

Participants must not be a beneficiary of government funded healthcare program (i.e. Medicare, Medicaid, etc.)

• Participants must not have a diagnosis of cancer within the past 5 years

Age Groups: Child, Adult, Older Adult
Study Population: 18-64 years of age male or female, no children, no incarcerated subjects
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2018-12-01 (Actual); Primary Completion 2021-12-01 (Estimated); Study Completion 2022-06-01 (Estimated)

PRIMARY OUTCOMES:
Patients' perspective through a patient led Survey of Health and quality of life via patient reported outcome measures using Visual analogue scale given at Baseline and follow up. Measuring effectiveness and quality of life from 0 to 10 | 36 months
  Collecting and analyzing quantitative and qualitative data to draw generalized outcome measures, on real world data. Data from the subject surveys will analyze and measure the effectiveness through a subjective observation via patients' perspective survey on footwash with or without oral medication and if it helped with the reduction or elimination of infections.

SECONDARY OUTCOMES:
Visual Analogue scales | 36 months
  By utilizing the Visual analogue scale from the patients' perspective will generate real world data

CONTACTS AND LOCATIONS:
Locations (1):
- DCABM, Land O' Lakes, Florida, United States

IPD SHARING:
Plan to Share IPD: No